CLINICAL TRIAL: NCT06335303
Title: A Randomised, Double-blind, Placebo-controlled, Dose-finding Study Evaluating Efficacy, Safety, and Tolerability of Different Oral Doses of BI 1819479 Over at Least 24 Weeks in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Study to Test Whether BI 1819479 Improves Lung Function in People With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1462-0004; 2023-508395-11-00 (Other: CTIS); U1111-1302-4283 (Other: WHO)
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BI 1819479 low dose treatment group (Experimental)
  Interventions: Drug: BI 1819479
- BI 1819479 medium dose treatment group (Experimental)
  Interventions: Drug: BI 1819479
- BI 1819479 high dose treatment group (Experimental)
  Interventions: Drug: BI 1819479
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 1819479

INTERVENTIONS:
Drug: BI 1819479 — BI 1819479
  Arms: BI 1819479 high dose treatment group; BI 1819479 low dose treatment group; BI 1819479 medium dose treatment group
Drug: Placebo matching BI 1819479 — Placebo matching BI 1819479
  Arms: Placebo group

SUMMARY:
This study is open to adults 40 years or older with idiopathic pulmonary fibrosis (IPF). People can join the study if they are not on any treatment for IPF are on stable treatment for at least 3 months before starting the study. The purpose of this study is to find out whether a medicine called BI 1819479 helps people with IPF. 3 different doses of BI 1819479 are tested in this study.

Participants are put into 4 groups by chance. Participants in 3 groups get different doses of BI 1819479. Participants in 1 group get placebo. Placebo tablets look like BI 1819479 tablets, but do not contain any medicine. Participants take the treatment for 6 months to 1 year. Participants are in the study for up to 1 year and 2 months. During this time, they visit the study site between 10 and 12 times and get up to 11 phone calls from the site staff.

At site visits doctors regularly perform breathing tests that measure how well the lungs are working. Researchers compare the results between participants who take BI 1819479 and placebo. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥40 years old at the time of signed informed consent.
2. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
3. Diagnosis of Idiopathic Pulmonary Fibrosis (IPF)
4. On stable treatment with nintedanib or pirfenidone for at least 12 weeks or not on treatment with either nintedanib or pirfenidone for at least 12 weeks
5. Forced Vital Capacity (FVC) ≥45% of predicted normal.
6. Diffusion capacity of the lung for carbon monoxide (DLCO) ≥25% of predicted normal corrected for hemoglobin (Hb).
7. Women of childbearing potential (WOCBP) must use highly effective methods of birth control with low user dependency and additional barrier contraception for male partners (use of condom) until end of follow-up period.
8. Male trial participants with WOCBP partners must use contraception (condom) to avoid exposure via seminal fluid. Female partners of male trial participants must use highly effective methods of contraception during treatment until end of follow-up period.

Exclusion Criteria:

1. Acute exacerbation of Idiopathic Pulmonary Fibrosis (IPF) within at least 12 weeks prior to screening and/or during the screening period (investigator-determined).
2. Treated with immunosuppressive medications (other than oral corticosteroids) or prednisone >15 mg/day or equivalent for respiratory or pulmonary reasons.
3. Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
4. The patient is currently enrolled in another investigational device or drug trial, or their Visit 1 occurs less than 30 days or 5 half-lives (whichever is longer) after completing a previous investigational device or drug trial or receiving other investigational treatments.
5. Patients with a significant disease or condition other than the IPF under study, which in the opinion of the investigator, may put the patient at risk because of participation, interfere with trial procedures, or cause concern regarding the patient's ability to participate in the trial or any medical condition which could lead to a life expectancy <12 months.
6. Relevant airways obstruction (pre-bronchodilator forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) <0.7).
7. In the opinion of the Investigator, other clinically significant pulmonary abnormalities.
8. Lower respiratory tract infection requiring treatment within 4 weeks prior to Visit 1 and/or during the screening period.

Further exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Annual rate of decline in Forced Vital Capacity (FVC) [milliLiter/year] | Up to 52 weeks

SECONDARY OUTCOMES:
Absolute change from baseline in FVC at Week 24 [in milliLiter] | At baseline and at week 24

CONTACTS AND LOCATIONS:
Locations (163):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Critical Care, Pulmonary and Sleep Associates, Lakewood, Colorado
  - Clinical Research Specialists LLC - Kissimmee, Kissimmee, Florida
  - SEC Clinical Research, Pensacola, Florida
  - The Iowa Clinic, PC, West Des Moines, Iowa
  - Advanced Pulmonary Research, Warren, Michigan
  - Memorial Hospital Gulfport, Gulfport, Mississippi
  - Coastal Carolina Health Care, P.A. Pulmonary and Sleep Medicine, New Bern, North Carolina
  - Southeastern Research Center-Winston Salem-69289, Winston-Salem, North Carolina
  - Clinical Research Associates of Central PA, DuBois, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Lowcountry Lung and Critical Care, Charleston, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Clinical Trials Center of Middle Tennessee, LLC, Franklin, Tennessee
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
- Argentina (5):
  - Centro de Investigaciones Metabolicas (CINME)-C.A.B.A-61553, C.a.b.a
  - Hospital Britanico de Buenos Aires, CABA
  - Centro de Investigación Clinica Belgrano, CABA
  - CEDIC - Centro de Investigacion Clinica, CABA
  - Consultorios Médicos del Buen Ayre, Capital Federal
- Australia (8):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Launceston Respiratory & Sleep Centre, Launceston, Tasmania
  - Lung Research Victoria, Footscray, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Institute for Respiratory Health, Nedlands, Western Australia
  - Macquarie University, Macquarie Park
- Austria (7):
  - Medical University of Graz State Hospital - University Hospital Graz, Graz
  - Krems University Hospital, Krems
  - Kepler Univ. Klinikum Linz, Linz
  - Hospital Elisabethinen Linz, Linz
  - Standort Penzing der Klinik Ottakring, Vienna
  - Clinic Floridsdorf, Vienna
  - Klinikum Wels - Grieskirchen GmbH, Wels
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHR de la Citadelle, Liège
- Brazil (7):
  - Serviços Medicos Respirar Sul Fluminense, Barra Mansa
  - Faculdade de Medicina de Botucatu - UNESP, Botucatu
  - Hospital das Clínicas da UFG - EBSERH, Goiânia
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Pesquisare, Santo André
  - COE Sao Jose dos Campos, São José dos Campos
  - Hospital Alemao Oswaldo Cruz, São Paulo
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Toronto General Hospital, Toronto, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
- China (14):
  - Beijing Chao-Yang Hospital, Beijing
  - The Second Xiangya Hospital Of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - People's Hospital of Sichuan Province, Chengdu
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Hangzhou First People's Hospital, Hangzhou
  - Zhejiang Hospital, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - Nanjing Drum Tower Hospital, Nanjing
  - China Shenyang Chest Hospital, Shenyang
  - Tianjin Medical University General Hospital, Tianjin
  - Tongji Hospital Affiliated Tongji Medical College Huazhong University of S & T, Wuhan
  - Affiliated Hospital, Xuzhou Medical college, Xuzhou
- Czechia (2):
  - University Thomayer´s Hospital, Prague
  - University Hospital Bulovka, Prague
- Denmark (2):
  - Rigshospitalet-København Ø-69883, København Ø
  - Odense University Hospital, Odense
- Finland (4):
  - HYKS Keuhkosairauksien tutkimusyksikkö, Helsinki
  - Oulun yliopistollinen keskussairaala, Oulu
  - Tampereen yliopistollinen sairaala, Tampere
  - TYKS, Turku
- France (8):
  - HOP d'Angers, Angers
  - HOP Avicenne, Bobigny
  - HOP Louis Pradel, Bron
  - HOP CHU Caen, Caen
  - INS Coeur Poumon, Lille
  - HOP Nord, Marseille
  - HOP Pasteur, Nice
  - HOP Pontchaillou, Rennes
- Germany (12):
  - Pneumologische Praxis Dr. Löh, Bad Homburg
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Caritas-Krankenhaus St. Maria gGmbH, Donaustauf
  - Klinikum Fulda gAG, Fulda
  - Universitätsmedizin Greifswald, Greifswald
  - Klinikum Region Hannover GmbH, Hanover
  - Lungenklinik Hemer, Hemer
  - Lungenfachklinik Immenhausen, Immenhausen
  - Klinikum Konstanz, Konstanz
  - Universität Leipzig, Leipzig
  - Klinikum der Universität München AÖR, München
- Greece (2):
  - Hospital of Heraklion (PAGNI), Crete
  - Univ. Gen. Hosp. of Ioannina, Ioannina
- University of Debrecen Clinical Centre, Debrecen, Hungary
- Italy (9):
  - A. O. Universitaria Careggi, Florence
  - Ospedale Colonnello D Avanzo, Foggia
  - Ospedale G.B. Morgagni, Forlì
  - Azienda Ospedaliera San Martino, Genova
  - Ospedale Classificato San Giuseppe, Milan
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Pol. Universitario Tor Vergata, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
- Japan (11):
  - Tosei General Hospital, Aichi, Seto
  - University of Fukui Hospital, Fukui, Yoshida-gun
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - Tokushima University Hospital, Tokushima, Tokushima
  - Kyorin University Hospital, Tokyo, Mitaka
  - Toho University Omori Medical Center, Tokyo, Ota-ku
  - National Center for Global Health and Medicine, Tokyo, Shinjuku-ku
- Malaysia (3):
  - Hospital Sultan Idris Shah Serdang, Kajang
  - Institut Perubatan Respiratori, Kuala Lumpur
  - Sarawak General Hospital, Kuching, Sarawak
- New Zealand (3):
  - Aotearoa Clinical Trials, Papatoetoe, Auckland
  - Waikato Hospital, Hamilton
  - Greenlane Clinical Centre, One Tree Hill, Auckland
- Norway (2):
  - Haukeland Universitetssykehus, Bergen
  - Akershus Universitetssykehus HF, Lørenskog
- Poland (2):
  - Clin.Hosp.Med.Univ.Marcinkowski in Poznan, Poznan
  - Alergopneuma Medical Center, Świdnik
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (8):
  - The Catholic University of Korea, Bucheon St.Mary's Hospital, Bucheon-si
  - Inje University Haeundae Paik Hospital, Busan
  - Seoul National University Bundang Hospital, Seongnam
  - Inje University Sanggye Paik Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Severance Hospital, Seoul
  - Soonchunhyang University Hospital Seoul, Seoul
  - Asan Medical Center, Seoul
- Spain (11):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital de Galdakao, Galdakao
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario De La Princesa, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocío, Seville
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - CTC Clinical Trial Consultants AB, Uppsala
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- Thailand (4):
  - Chulalongkorn Hospital, Bangkok
  - Srinagarind Hospital, Khon Kaen
  - Ramathibodi Hospital, Ratchathewi
  - Songklanagarind Hospital, Thailand
- United Kingdom (8):
  - Heartlands Hospital, Birmingham
  - Castle Hill Hospital, Cottingham, Hull
  - Royal Devon and Exeter Hospital, Wonford, Exeter
  - Royal Lancaster Infirmary, Lancaster
  - St James's University Hospital, Leeds
  - Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com